CLINICAL TRIAL: NCT01822418
Title: Agomelatine Treatment of Major Depressive Episodes in the Course of Schizophrenic Psychoses (AGOPSYCH)
Brief Title: Agomelatine Treatment of Depression in Schizophrenia (AGOPSYCH)
Acronym: AGOPSYCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01112012
Record Dates: First submitted 2013-03-11; First posted 2013-04-02 (Estimated); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Delusional Disorder
Keywords: Schizophrenia; Depression; Cognition; Agomelatine; Antidepressant
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid; Depression | interventions — agomelatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Open-label treatment with agomelatine 25 mg/day (or 50 mg/day after week 3).
  Interventions: Drug: agomelatine

INTERVENTIONS:
Drug: agomelatine — Augmentation of antipsychotic therapy with 25 to 50 mg agomelatine as a single oral dosage per day
  Other Names: Valdoxan

SUMMARY:
Major depressive episodes (MDEs) occur frequently during the course of psychotic disorders, and several antidepressive agents have been successfully applied. The new melatonergic antidepressant agomelatine (AGO) appears promising for the treatment of MDEs in schizophrenia for several reasons. The investigators plan to test the efficacy and tolerability of AGO for antidepressive treatment in schizophrenia. For this task, the investigators plan to enrol 27 schizophrenic patients into an open, single-armed, prospective clinical trial with agomelatine.

DETAILED DESCRIPTION:
Major depressive episodes (MDEs) occur frequently during the course of psychotic disorders, and several antidepressive agents have been successfully applied. The new melatonergic antidepressant agomelatine (AGO) appears promising for the treatment of MDEs in schizophrenia for several reasons: 1. AGO provides a unique pharmacological profile by combining antidepressive potency, sleep regulation and enhancement of frontocortical dopaminergic activity by 5-HT-2C-blockade. 2. AGO might exert favourable effects on cognition. 3. While pharmacokinetic interactions are generally possible, major influences on antipsychotic substances are unlikely due to metabolism by cytochrome isoenzymes CYP1A2 and CYP2C9/19. 4. AGO is characterized by a favourable range of adverse events (AE) which do not overlap with typical antipsychotic AEs such as weight gain and sexual dysfunction. Thus, the risk of additive effects seems to be small. The investigators plan to enroll 27 schizophrenic patients into an open, single-armed, prospective clinical trial with agomelatine. As predefined primary and secondary endpoints, we are going to investigate whether AGO is able to improve MDE severity, sleep quality, general and psychosocial functioning as well as cognitive function in schizophrenia without detrimental effects on the psychotic syndrome. Moreover, we intend to monitor for pharmacokinetic interactions. The results obtained will allow designing future randomized and controlled clinical trials in order to improve the range of therapeutic options for affective and cognitive deficits in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years.
2. Presence of an MDE according to ICD-10 criteria (HAMD17 ≥ 18 or CDSS-Score ≥ 8 points).
3. Lifetime diagnosis of schizophrenia-spectrum disorder according to ICD-10 (F 20, F22, F23, F25).
4. Partial remission of psychotic positive symptoms (PANSS positive subscore ≤ 15 points).
5. Stable antipsychotic medication for at least 2 weeks (tolerable quantitative changes of daily dosage ≤ 25%).
6. The patient is able to give an informed consent. In case of legal guardianship, the custodian will have to agree to the patient's participation.

Exclusion Criteria:

1. Contraindications against AGO treatment
2. Insufficient contraception in women of childbearing potential when sexually active.
3. Gravidity or breastfeeding.
4. Addiction to alcohol
5. Current abuse of THC and other illegal substances according to ICD-10
6. Dementia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Antidepressive efficacy | 6 weeks
  Comparison of MDE severity before and after six weeks of treatment with AGO. In order to assess the treatment success, means of HAM-D17 and CDSS scores at both baseline and week 6 will be compared within the efficacy sample (at least one application of AGO, LOCF). The primary endpoint will be tested with a two-sided student's t-test at a level of statistical significance of ≤.05.

SECONDARY OUTCOMES:
Secondary efficacy measures: Response rates | 6 weeks and 3 months
  We will determine the percentage of responses (decrease of HAMD by at least 50 %)
Secondary efficacy measures: Long-term efficacy | 6 weeks and 3 months
  After 12 weeks of treatment we plan to compare means of HAMD and CDSS with baseline data.
Secondary efficacy measures: Psychosocial functioning | 6 weeks and 3 months
  During treatment psychosocial functioning might improve. We plan to compare means of PSP scale assessed after 6 weeks and 3 months with baseline data.
Secondary tolerability and safety measures: Psychotic symptoms | 6 weeks and 3 months
  The stability of the psychotic syndrome during treatment with AGO will be evaluated comparing means of PANSS after 6 weeks and 3 months with baseline.
Secondary tolerability and safety measures: General tolerability | 6 weeks and 3 months
  The general tolerability measures include the exploration and documentation of adverse events.
Secondary tolerability and safety measures: Pharmacokinetic interactions between AGO and antipsychotic agents | 6 weeks and 3 months
  Effects of AGO treatment on serum drug levels of antipsychotic agents will be evaluated by comparing the SDLs at baseline with values obtained after 6 weeks and 3 months.
Secondary efficacy measures: Remission rates | 6 weeks and 3 months
  We will determine the percentage of remissions (decrease of HAMD below 8)
Secondary efficacy measures: Cognitive functioning | 3 months
  During treatment neurocognitive deficits might improve. We plan to compare means in the MCCB assessed after 3 months with baseline data.

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Zink, MD, Principal Investigator — Central Institute of Mental Health, Department of Psychiatry and Psychotherapy
Locations (1):
- Central Institute of Mental Health, Mannheim, Baden-Wurttemberg, Germany

REFERENCES:
- See also: Central Institute of Mental Health. Non-profit University hospital — https://www.zi-mannheim.de